CLINICAL TRIAL: NCT03028194
Title: Effects of Postpartum Uterine Curettage in the Recovery From Preeclampsia/Eclampsia: A Randomized, Controlled Trial
Brief Title: Postpartum Uterine Curettage in the Recovery From Preeclampsia/Eclampsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Head of the Research Department, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2014-06
Record Dates: First submitted 2017-01-18; First posted 2017-01-23 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Pre-Eclampsia; Eclampsia
Keywords: Pre-eclampsia; Eclampsia; Postpartum uterine curettage
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia | interventions — Curettage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Curettage (Experimental): Postpartum uterine curettage performed immediately after delivery of the placenta.
  Interventions: Procedure: Curettage
- Placebo (Placebo Comparator): No procedure performed after delivery of the placenta.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Curettage — Postpartum uterine curettage with a sharp curette # 14 or #16, immediately after delivery of the placenta.
  Arms: Curettage
Procedure: Placebo — No procedure after delivery of the placenta
  Arms: Placebo

SUMMARY:
Use of Postpartum uterine curettage in reducing hospitalization time or in improving the clinical evolution of the patient with preeclampsia/eclampsia.

DETAILED DESCRIPTION:
To evaluate if postpartum uterine curettage improved the clinical and laboratory parameters in patients with preeclampsia or eclampsia.

A total of 442 patients with preeclampsia/eclampsia were randomized to postpartum curettage (223) or no procedure (219). Systolic and diastolic blood pressure were recorded and analyzed at hours 6, 12, 24 and 48. Also, several laboratory values and diuresis were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24 weeks or more.
* Preeclampsia/eclampsia

Exclusion Criteria:

* Epilepsy or seizures previous to pregnancy.
* Renal disease
* Heart disease
* Liver disease

Ages: 15 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 442 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-12-11 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 6 hours
  Arterial blood pressure
Systolic and diastolic blood pressure | 12 hours
  Arterial blood pressure
Systolic and diastolic blood pressure | 24 hours
  Arterial blood pressure
Systolic and diastolic blood pressure | 48 hours
  Arterial Blood pressure

SECONDARY OUTCOMES:
Laboratory results (hypertensive disorder profile: hemoglobin, hematocrit, platelets, renal or liver function tests). | 6 hours
  Number of patients with an abnormal laboratory value
Laboratory results (hypertensive disorder profile: hemoglobin, hematocrit, platelets, renal or liver function tests). | 12 hours
  Number of patients with an abnormal laboratory value
Laboratory results (hypertensive disorder profile: hemoglobin, hematocrit, platelets, renal or liver function tests). | 24 hours
  Number of patients with an abnormal laboratory value
Laboratory results (hypertensive disorder profile: hemoglobin, hematocrit, platelets, renal or liver function tests). | 48 hours
  Number of patients with an abnormal laboratory value
Seizures | 48 hours
  Number of participants with the development of seizures after birth.

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, MD, Study Chair — Saint Thomas Hospital, Panama
Locations (2):
- Panama (2):
  - Saint Thomas H, Panama City, Provincia de Panamá
  - Saint Thomas Maternity Hospital, Panama City, Provincia de Panamá

IPD SHARING:
Plan to Share IPD: No